CLINICAL TRIAL: NCT00702754
Title: An Open Label Safety and Immunogenicity Study of MYOBLOC (Neurobloc; Botulinum Toxin Type B) Injectable Solution in Patients With Cervical Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solstice Neurosciences (Industry)
Responsible Party: Sponsor
Organization: USWM, LLC (dba US WorldMeds) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 401CDNA; 401CDNA
Record Dates: First submitted 2008-06-12; First posted 2008-06-20 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — rimabotulinumtoxinB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Botulinum Toxin Type B — Eligible patients could receive injections of MYOBLOC once every 12 weeks. Total Dose could range from 5,000 Units up to 25,000 Units.
  Other Names: MYOBLOC

SUMMARY:
Five hundred patients with a confirmed clinical diagnosis of Cervical Dystonia (CD)are planned for enrollment into this open label study. These patients will be Type B toxin naive patients with CD. During this study patients will receive repeat injections of MYOBLOC when deemed appropriate by the Investigator. However, it will be recommended that injections occur not more frequently than every 12 weeks. Total duration of exposure to MYOBLOC will be targeted for at least two years, with potential exposure for up to 7 years in patients with earliest enrollment

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* body weight of at least 46 kilograms
* History of Cervical Dystonia of at least one year's duration who in the opinion of the Investigator requires treatment

Exclusion Criteria:

* Inability to give informed consent
* Patient who has been previously treated with botulinum Toxin Type B
* Patient who has received a Botulinum toxin Type A injection in the last 12 weeks.
* History of phenol injections involving the neck or shoulder region in the last 12 months.
* Patients with neck contractures or cervical spine disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2001-06; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 500 subjects were recruited from 36 centers in North America.
Pre-assignment Details: Subjects had to be Botulinum Toxin Type B naive and could not have received a Botulinum Toxin Type A treatment within 12 weeks of enrollment.
Groups:
- MYOBLOC Open Label Treatment: All patients meeting enrollment criteria received open-label MYOBLOC. Patients were eligible for repeat injections approximately every 12 weeks.
Period: MYOBLOC Treatment Session 1 (Time 0)
Arm/Group | MYOBLOC Open Label Treatment
Started | 502
Completed | 495 (Approximately 70% of subjects completed at least 2 years of treatment.)
Not Completed | 7
Period: MYOBLOC Treatment Session 2 (App 12 Wks)
Arm/Group | MYOBLOC Open Label Treatment
Started | 495
Completed | 475
Not Completed | 20
Period: MYOBLOC Treatment Session 3 (App 24 Wks)
Arm/Group | MYOBLOC Open Label Treatment
Started | 475
Completed | 450
Not Completed | 25
Period: MYOBLOC Treatment Session 4 (App 36 Wks)
Arm/Group | MYOBLOC Open Label Treatment
Started | 450
Completed | 428
Not Completed | 22
Period: MYOBLOC Treatment Session 5 (App 48 Wks)
Arm/Group | MYOBLOC Open Label Treatment
Started | 428
Completed | 396
Not Completed | 32
Period: MYOBLOC Treatment Session 6 (App 60 Wks)
Arm/Group | MYOBLOC Open Label Treatment
Started | 396
Completed | 377
Not Completed | 19
Period: MYOBLOC Treatment Session 7 (App 72 Wks)
Arm/Group | MYOBLOC Open Label Treatment
Started | 377
Completed | 353
Not Completed | 24
Period: MYOBLOC Treatment Session 8 (App 84 Wks)
Arm/Group | MYOBLOC Open Label Treatment
Started | 353
Completed | 329
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 502
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 419
  >=65 years | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341
  Male | 161
Region of Enrollment [Number; unit: participants]
  North America | 502

OUTCOME MEASURES:

1. Primary Outcome: Treatment Assessment Scale (TAS), 4 Wks Post-injection Compared to Baseline (Time 0), Rating of Cervical Dystonia Symptoms
Description: 7 point rating scale (-3 = significantly worse, 0 = no change, +3 = significantly better. Comparison at Wk 4 to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 1 - Time 0, 4 weeks post-injection compared to baseline
Population: Safety Population/Intent to Treat
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 495
points on a scale | 0.9 (0.1) [-3 to 3]

2. Secondary Outcome: Treatment Assessment Scale (TAS), Approx Wk 12 + 4 Wks Post-Injection Compared to Baseline. Rating of Cervical Dystonia Symptoms
Description: 7 point rating scale (-3=significantly worse, 0=no change, +3=significantly better), comparison of Wk 12 + 4, compared to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 2 (12 wks) - 4 weeks post-injection compared to baseline
Population: safety population/Intent to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 475
points on a scale | 1.3 (0.1)

3. Secondary Outcome: Treatment Assessment Scale (TAS), Approx Wk 24 + 4 Wks Post-injection Compared to Baseline. Rating of Cervical Dystonia Symptoms
Description: 7 point scale (-3=significantly worse, 0=no change, +3=significantly better). Comparison of Wk 24 + 4, compared to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 3 (24 Wks) - 4 weeks post-injection compared to baseline
Population: safety population/Intent to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 450
points on a scale | 1.5 (0.1)

4. Secondary Outcome: Treatment Assessment Scale (TAS), Approx Wk 36 + 4 Wks Post-injection Compared to Baseline. Rating of Cervical Dystonia Symptoms
Description: 7 point scale (-3=significantly worse, 0=no change, +3=significantly better). Comparison of Wk 36 + 4, compared to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 4 (36 Wks) - 4 weeks post-injection compared to baseline
Population: safety population/Intent to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 428
points on a scale | 1.4 (0.1)

5. Secondary Outcome: Treatment Assessment Scale (TAS), Approx Wk 48 + 4 Wks Post-injection Compared to Baseline. Rating of Cervical Dystonia Symptoms
Description: 7 point scale (-3=significantly worse, 0=no change, +3=significantly better). Comparison of Wk 48 + 4, compared to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 5 (48 Wks) - 4 weeks post-injection compared to baseline
Population: Safety Population/Intent to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 396
points on a scale | 1.5 (0.1) [-3 to 3]

6. Secondary Outcome: Treatment Assessment Scale (TAS), Approx Wk 60 + 4 Wks Post-injection Compared to Baseline. Rating of Cervical Dystonia Symptoms
Description: 7 point scale (-3=significantly worse, 0=no change, +3=significantly better). comparison Wk 60 + 4, compared to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 6 (60 Wks) - 4 weeks post-injection compared to baseline
Population: Safety Population/Intent to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 377
points on a scale | 1.4 (0.1)

7. Secondary Outcome: Treatment Assessment Scale (TAS), Approx Wk 72 + 4 Wks Post-injection Compared to Baseline. Rating of Cervical Dystonia Symptoms
Description: 7 point scale (-3=significantly worse, 0=no change, +3=significantly better). Comparison Wk 72 + 4, compared to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 7 (72 Wks) - 4 weeks post-injection compared to baseline
Population: Safety Population/Intent to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 353
points on a scale | 1.5 (0.1)

8. Secondary Outcome: Treatment Assessment Scale (TAS), Approx Wk 84 + 4 Wks Post-injection Compared to Baseline. Rating of Cervical Dystonia Symptoms
Description: 7 point scale (-3=significantly worse, 0=no change, +3=significantly better). Comparison Wk 84 + 4, compared to baseline. Rating of Cervical Dystonia Symptoms
Time Frame: Session 8 (84 Wks) - 4 weeks post-injection compared to baseline
Population: Safety Population/Intent to Treat
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | MYOBLOC Open Label Treatment
Number analyzed (Participants) | 329
points on a scale | 1.4 (0.1)

ADVERSE EVENTS:
Arm/Group | MYOBLOC Open Label Treatment
Serious Adverse Events (participants affected / at risk) | 133
Other Adverse Events (participants affected / at risk) | 494
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | MYOBLOC Open Label Treatment
Acute Coronary Syndrome (Cardiac disorders) | 8/502 (8)
Acute Myocardial Infarction (Cardiac disorders) | 1/502 (1)
Angina (Cardiac disorders) | 1/502 (1)
Atrial Fibrillation (Cardiac disorders) | 3/502 (3)
AV Block 2nd Degree (Cardiac disorders) | 1/502 (1)
Coronary Artery Occlusion (Cardiac disorders) | 1/502 (1)
Bradycardia (Cardiac disorders) | 1/502 (1)
Myocardial infarction (Cardiac disorders) | 2/502 (2)
Palpitations (Cardiac disorders) | 1/502 (1)
Pericardial effusion (Cardiac disorders) | 1/502 (1)
sinus bradycardia (Cardiac disorders) | 1/502 (1)
tachycardia (Cardiac disorders) | 1/502 (1)
vertigo (Ear and labyrinth disorders) | 1/502 (1)
adrenal insufficiency (Endocrine disorders) | 1/502 (1)
eye haemorrhage (Eye disorders) | 1/502 (1)
abdominal adhesions (Gastrointestinal disorders) | 1/502 (1)
abdominal pain (Gastrointestinal disorders) | 2/502 (2)
appendicitis (Gastrointestinal disorders) | 1/502 (1)
celiac disease (Gastrointestinal disorders) | 1/502 (1)
constipation (Gastrointestinal disorders) | 1/502 (1)
diarrhea (Gastrointestinal disorders) | 1/502 (1)
diverticulum (Gastrointestinal disorders) | 1/502 (1)
dysphagia (Gastrointestinal disorders) | 1/502 (1)
GI hemorrhage (Gastrointestinal disorders) | 3/502 (3)
GI Reflux disease (Gastrointestinal disorders) | 1/502 (1)
inguinal hernia (Gastrointestinal disorders) | 1/502 (1)
inguinal hernia obsstructive (Gastrointestinal disorders) | 1/502 (1)
nausea (Gastrointestinal disorders) | 1/502 (1)
pancreatitis (Gastrointestinal disorders) | 1/502 (1)
small intestine obstruction (Gastrointestinal disorders) | 1/502 (1)
upper GI hemorrhage (Gastrointestinal disorders) | 1/502 (1)
vomiting (Gastrointestinal disorders) | 2/502 (2)
chest discomfort (General disorders) | 1/502 (1)
chest pain (General disorders) | 4/502 (4)
facial pain (General disorders) | 1/502 (1)
non cardiac chest pain (General disorders) | 1/502 (1)
pain (General disorders) | 1/502 (1)
bile duct stone (Hepatobiliary disorders) | 1/502 (1)
cholecystitis (Hepatobiliary disorders) | 1/502 (1)
cholecystitis acute (Hepatobiliary disorders) | 1/502 (1)
cholelithiasis (Hepatobiliary disorders) | 4/502 (4)
hepatorenal syndrome (Hepatobiliary disorders) | 1/502 (1)
jaundice (Hepatobiliary disorders) | 1/502 (1)
hypersensitivity (Immune system disorders) | 1/502 (1)
abdominal abscess (Infections and infestations) | 1/502 (1)
appendicitis (Infections and infestations) | 1/502 (1)
arthritis infective (Infections and infestations) | 1/502 (1)
bartholin abscess (Infections and infestations) | 1/502 (1)
GI norwalk virus (Infections and infestations) | 1/502 (1)
GI viral (Infections and infestations) | 1/502 (1)
haemophilis infection (Infections and infestations) | 1/502 (1)
pelvic abscess (Infections and infestations) | 1/502 (1)
pneumonia (Infections and infestations) | 2/502 (2)
post operative abscess (Infections and infestations) | 1/502 (1)
pyelonephritis (Infections and infestations) | 1/502 (1)
sinusitis (Infections and infestations) | 1/502 (1)
Upper Respiratory Infection (URI) (Infections and infestations) | 1/502 (1)
Urinary Tract Infection (UTI) (Infections and infestations) | 1/502 (1)
vaginal cellulitis (Infections and infestations) | 1/502 (1)
accidental overdose (Injury, poisoning and procedural complications) | 1/502 (1)
brain contusion (Injury, poisoning and procedural complications) | 1/502 (1)
clavicle fracture (Injury, poisoning and procedural complications) | 1/502 (1)
drug toxicitiy (Infections and infestations) | 1/502 (1)
fall (Injury, poisoning and procedural complications) | 1/502 (1)
hip fracture (Injury, poisoning and procedural complications) | 3/502 (3)
incisional hernia (Injury, poisoning and procedural complications) | 2/502 (2)
medication error (Injury, poisoning and procedural complications) | 1/502 (1)
multiple fractures (Injury, poisoning and procedural complications) | 1/502 (1)
overdose (Injury, poisoning and procedural complications) | 20/502 (20)
post procedural nausea (Injury, poisoning and procedural complications) | 1/502 (1)
post pocedural vomiting (Injury, poisoning and procedural complications) | 1/502 (1)
post operative ileus (Injury, poisoning and procedural complications) | 1/502 (1)
road traffic accident (Injury, poisoning and procedural complications) | 4/502 (4)
subdural hematoma (Injury, poisoning and procedural complications) | 1/502 (1)
upper limb fracture (Injury, poisoning and procedural complications) | 1/502 (1)
oxygen saturation decrease (Investigations) | 1/502 (1)
dehydration (Metabolism and nutrition disorders) | 3/502 (3)
hyperglycemia (Metabolism and nutrition disorders) | 1/502 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1/502 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1/502 (1)
back disorder (Musculoskeletal and connective tissue disorders) | 1/502 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1/502 (1)
intervebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2/502 (2)
intervebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2/502 (2)
muscle spasm (Musculoskeletal and connective tissue disorders) | 1/502 (1)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/502 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 2/502 (2)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1/502 (1)
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2/502 (2)
torticollis (Musculoskeletal and connective tissue disorders) | 7/502 (7)
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/502 (4)
basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5/502 (5)
keratocanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/502 (2)
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/502 (2)
squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/502 (1)
Cerebrovascular Accident (CVA) (Nervous system disorders) | 3/502 (3)
cervical myelopathy (Nervous system disorders) | 2/502 (2)
convulsion (Nervous system disorders) | 1/502 (1)
Dementia (Nervous system disorders) | 1/502 (1)
Dizziness (Nervous system disorders) | 2/502 (2)
dystonia (Nervous system disorders) | 1/502 (1)
epilepsy (Nervous system disorders) | 1/502 (1)
intracranial aneurysm (Nervous system disorders) | 1/502 (1)
mutiple sclerosis (Nervous system disorders) | 2/502 (2)
syncope (Nervous system disorders) | 1/502 (1)
vertebrobasilar insufficiency (Nervous system disorders) | 1/502 (1)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 2/502 (2)
anxiety (Psychiatric disorders) | 1/502 (1)
confusional state (Psychiatric disorders) | 1/502 (1)
depression (Psychiatric disorders) | 3/502 (3)
dissociative identity disorder (Psychiatric disorders) | 1/502 (1)
major depression (Psychiatric disorders) | 1/502 (1)
suicidal ideation (Psychiatric disorders) | 3/502 (3)
bladder prolapse (Renal and urinary disorders) | 1/502 (1)
renal failure acute (Renal and urinary disorders) | 1/502 (1)
stress incontinence (Renal and urinary disorders) | 1/502 (1)
cystocele (Reproductive system and breast disorders) | 1/502 (1)
endometriosis (Reproductive system and breast disorders) | 1/502 (1)
menorrhagia (Reproductive system and breast disorders) | 1/502 (1)
ovarian cyst (Reproductive system and breast disorders) | 1/502 (1)
ovarian cyst rupture (Reproductive system and breast disorders) | 1/502 (1)
pelvic peritoneal adhesions (Reproductive system and breast disorders) | 1/502 (1)
rectocele (Reproductive system and breast disorders) | 1/502 (1)
atelectasis (Reproductive system and breast disorders) | 2/502 (2)
choking (Respiratory, thoracic and mediastinal disorders) | 1/502 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2/502 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2/502 (2)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/502 (2)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1/502 (1)
sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1/502 (1)
blood pressure fluctuation (Vascular disorders) | 1/502 (1)
deep vein thrombosis (Vascular disorders) | 1/502 (1)
haemotoma (Vascular disorders) | 1/502 (1)
hypertension (Vascular disorders) | 3/502 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | MYOBLOC Open Label Treatment
Palpitations (Cardiac disorders) | 11/502 (11)
vertigo (Ear and labyrinth disorders) | 18/502 (18)
hypothyroidism (Endocrine disorders) | 10/502 (10)
cataract (Eye disorders) | 10/502 (10)
conjunctivitis (Eye disorders) | 11/502 (11)
dry eye (Eye disorders) | 10/502 (10)
vision blurred (Eye disorders) | 12/502 (12)
abdominal pain (Gastrointestinal disorders) | 29/502 (29)
abdominal pain upper (Gastrointestinal disorders) | 15/502 (15)
constipation (Gastrointestinal disorders) | 43/502 (43)
diarrhea (Gastrointestinal disorders) | 48/502 (48)
dry mouth (Gastrointestinal disorders) | 348/502 (348)
dyspepsia (Gastrointestinal disorders) | 48/502 (48)
dysphagia (Gastrointestinal disorders) | 203/502 (203)
GERD (Gastrointestinal disorders) | 42/502 (42)
nausea (Gastrointestinal disorders) | 72/502 (72)
toothache (Gastrointestinal disorders) | 10/502 (10)
vomiting (Gastrointestinal disorders) | 30/502 (30)
asthenia (General disorders) | 12/502 (12)
chest pain (General disorders) | 28/502 (28)
fatigue (General disorders) | 51/502 (51)
influenza like illness (General disorders) | 25/502 (25)
injection site pain (General disorders) | 114/502 (114)
injection site reaction (General disorders) | 15/502 (15)
edema peripheral (General disorders) | 26/502 (26)
pyrexia (General disorders) | 12/502 (12)
bronchitis (Infections and infestations) | 50/502 (50)
cystitis (Infections and infestations) | 18/502 (18)
ear infection (Infections and infestations) | 10/502 (10)
fungal infection (Infections and infestations) | 10/502 (10)
GI viral (Infections and infestations) | 24/502 (24)
herpes zoster (Infections and infestations) | 10/502 (10)
influenza (Infections and infestations) | 84/502 (84)
nasopharyngitis (Infections and infestations) | 110/502 (110)
otitis media (Infections and infestations) | 18/502 (18)
pneumonia (Infections and infestations) | 10/502 (10)
sinusitis (Infections and infestations) | 68/502 (68)
tooth abscess (Infections and infestations) | 14/502 (14)
Upper Respiratory Infection (Infections and infestations) | 70/502 (70)
joint sprain (Injury, poisoning and procedural complications) | 15/502 (15)
muscle sprain (Injury, poisoning and procedural complications) | 10/502 (10)
overdose (Injury, poisoning and procedural complications) | 20/502 (20)
procedural pain (Injury, poisoning and procedural complications) | 25/502 (25)
road traffic accident (Injury, poisoning and procedural complications) | 16/502 (16)
blood cholesterol increased (Investigations) | 11/502 (11)
hypercholesterolemia (Metabolism and nutrition disorders) | 22/502 (22)
arthralgia (Musculoskeletal and connective tissue disorders) | 61/502 (61)
arthritis (Musculoskeletal and connective tissue disorders) | 18/502 (18)
back pain (Musculoskeletal and connective tissue disorders) | 77/502 (77)
intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 12/502 (12)
interverterbral disc protrusion (Musculoskeletal and connective tissue disorders) | 11/502 (11)
muscle spasm (Musculoskeletal and connective tissue disorders) | 77/502 (77)
muscle tightness (Musculoskeletal and connective tissue disorders) | 13/502 (13)
muscle weakness (Musculoskeletal and connective tissue disorders) | 41/502 (41)
musculoskeletal weakness (Musculoskeletal and connective tissue disorders) | 20/502 (20)
myalgia (Musculoskeletal and connective tissue disorders) | 25/502 (25)
neck pain (Musculoskeletal and connective tissue disorders) | 32/502 (32)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 18/502 (18)
pain in extremity (Musculoskeletal and connective tissue disorders) | 56/502 (56)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 15/502 (15)
shoulder pain (Musculoskeletal and connective tissue disorders) | 29/502 (29)
tendonitis (Musculoskeletal and connective tissue disorders) | 15/502 (15)
torticollis (Musculoskeletal and connective tissue disorders) | 170/502 (170)
balance disorder (Nervous system disorders) | 13/502 (13)
carpal tunnel syndrome (Nervous system disorders) | 11/502 (11)
dizziness (Nervous system disorders) | 68/502 (68)
head titubation (Nervous system disorders) | 29/502 (29)
headache (Nervous system disorders) | 117/502 (117)
hypoaesthesia (Nervous system disorders) | 46/502 (46)
Migraine (Nervous system disorders) | 22/502 (22)
paraesthesia (Nervous system disorders) | 31/502 (31)
Somnolence (Nervous system disorders) | 19/502 (19)
syncope (Nervous system disorders) | 12/502 (12)
tremor (Nervous system disorders) | 33/502 (33)
anxiety (Psychiatric disorders) | 36/502 (36)
depression (Psychiatric disorders) | 67/502 (67)
insomnia (Psychiatric disorders) | 46/502 (46)
stress (Psychiatric disorders) | 12/502 (12)
choking (Respiratory, thoracic and mediastinal disorders) | 14/502 (14)
cough (Respiratory, thoracic and mediastinal disorders) | 51/502 (51)
dry throat (Respiratory, thoracic and mediastinal disorders) | 15/502 (15)
dysphonia (Respiratory, thoracic and mediastinal disorders) | 10/502 (10)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 19/502 (19)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17/502 (17)
pharangolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 36/502 (36)
pruritis (Skin and subcutaneous tissue disorders) | 10/502 (10)
rash (Skin and subcutaneous tissue disorders) | 31/502 (31)
hypertension (Vascular disorders) | 43/502 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual PI can disclose results until after a group manuscript is published.